CLINICAL TRIAL: NCT07151118
Title: Role of Circulating Tumor DNA (ctDNA) in Genetic Profiling and Clinical Outcomes for Advanced Biliary Tract Cancer (BTC) Patients - Prospective, Observational, Epidemiology Study
Brief Title: ctDNA in Genetic Profiling and Clinical Outcomes of Advanced Biliary Tract Cancer
Status: Not yet recruiting | Type: Observational
Sponsor: CHA University (Other)
Collaborators: Handok Inc. (Industry)
Responsible Party: Principal Investigator, Hong Jae Chon, Principal Investigator, CHA University
Other Study IDs: CHAMC2025-03-041
Record Dates: First submitted 2025-08-20; First posted 2025-09-03 (Actual); Last update posted 2025-09-09 (Actual); Status verified 2025-09

CONDITIONS: Biliary Tract Cancer
Keywords: Biliary Tract Cancer; Biomarker; IDH1 mutation; FGFR2 fusion; Circulating Tumor DNA (ctDNA); Biomarker Analysis
MeSH Terms: conditions — Biliary Tract Neoplasms | interventions — Blood Specimen Collection; Liquid Biopsy

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Blood
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Advanced Biliary Tract Cancer Patients: Patients with histologically confirmed advanced or metastatic biliary tract cancer (intrahepatic cholangiocarcinoma, extrahepatic cholangiocarcinoma, or gallbladder cancer). Participants will provide blood samples for circulating tumor DNA (ctDNA) analysis before systemic therapy or prior to subsequent treatment.
  Interventions: Other: Blood Sampling for ctDNA Analysis

INTERVENTIONS:
Other: Blood Sampling for ctDNA Analysis — Approximately 20 mL of peripheral blood will be collected from patients with advanced biliary tract cancer. Samples will be obtained prior to systemic therapy initiation (in about two-thirds of patients) or prior to subsequent therapy (in about one-third of patients). Additional blood draws may be performed at progression in patients with FGFR2 fusion, IDH1 mutation, or HER2 amplification. Collected samples will be centrally analyzed for genomic alterations using ctDNA profiling.
  Other Names: Liquid Biopsy; Plasma Collection

SUMMARY:
This prospective, multicenter, observational study aims to evaluate the role of circulating tumor DNA (ctDNA) in advanced or metastatic biliary tract cancer (BTC) patients in Korea. Tissue-based genomic profiling is often limited due to the anatomical challenges of tumor biopsy and insufficient DNA quality. ctDNA analysis offers a minimally invasive alternative for identifying actionable genetic alterations, including Fibroblast Growth Factor Receptor 2 (FGFR2) fusions, Isocitrate Dehydrogenase 1 (IDH1) mutations, and Human Epidermal Growth Factor Receptor 2 (HER2) amplifications. The study will recruit 100 patients across 11 institutions and assess the concordance between ctDNA and tissue genomic profiling, as well as the clinical relevance of ctDNA in predicting treatment outcomes and prognosis.

DETAILED DESCRIPTION:
Biliary tract cancer (BTC) is a heterogeneous and aggressive malignancy with poor prognosis, especially in advanced or metastatic stages where surgical resection is not feasible. The current standard first-line therapy with gemcitabine and cisplatin provides limited survival benefit, with median overall survival around 11-12 months. Targeted therapies, such as FGFR inhibitors for FGFR2 fusions and IDH1 inhibitors, as well as immune checkpoint inhibitors, have improved outcomes in subsets of patients. However, tumor tissue acquisition remains challenging in BTC, limiting the ability to perform comprehensive genomic profiling.

Circulating tumor DNA (ctDNA) has emerged as a promising biomarker for molecular profiling, treatment monitoring, and prognosis assessment. Prior studies demonstrated acceptable concordance between ctDNA-based and tissue-based next-generation sequencing, particularly for FGFR2 fusions, and highlighted the potential of ctDNA in identifying additional genomic alterations not detected in tissue samples.

This prospective study will enroll 100 Korean patients with advanced or metastatic BTC from 11 hospitals. Approximately two-thirds of patients will provide blood samples prior to first-line systemic therapy, while one-third will provide samples before subsequent therapy. Additional blood draws will be performed at progression in patients harboring FGFR2 fusion, IDH1 mutation, or HER2 amplification. Collected samples will be analyzed by a central laboratory (SCL Healthcare, a precision medicine service provider specializing in biomarker-based diagnostics).

The primary objective is to evaluate the frequency of actionable genomic alterations, especially FGFR2 fusions, detected by ctDNA in advanced BTC patients. Secondary objectives include:

* Assessing the concordance between ctDNA and tissue genomic profiling
* Evaluating the proportion of patients who received targeted therapy based on ctDNA results (e.g., pemigatinib [Pemazyre®])
* Exploring associations between ctDNA maximum variant allele frequency (max VAF) and survival outcomes
* Identifying potential resistance mechanisms and clonal evolution during targeted therapy

This study is expected to provide robust evidence for the clinical utility of ctDNA in BTC and contribute to the establishment of precision medicine approaches, potentially supporting future guideline development and regulatory approval of ctDNA assays in Korea and globally.

ELIGIBILITY:
Inclusion Criteria:

* Histologically confirmed advanced or metastatic biliary tract cancer (including intrahepatic cholangiocarcinoma, extrahepatic cholangiocarcinoma, and gallbladder carcinoma)
* Patients meeting one of the following conditions:

  * Prior to initiation of first-line systemic therapy
  * Patients who previously received systemic therapy and are able to provide a blood sample prior to initiation of subsequent therapy
* Age ≥ 19 years at the time of enrollment
* Willingness and ability to provide blood samples for ctDNA analysis

Exclusion Criteria:

* Refusal to provide blood samples for ctDNA testing
* Inability to provide written informed consent

Min Age: 19 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Korean patients with advanced or metastatic biliary tract cancer (intrahepatic, extrahepatic, or gallbladder carcinoma), enrolled for ctDNA-based genetic profiling prior to systemic therapy or before subsequent treatment initiation.
Sampling Method: Non-Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2025-09-01 (Estimated); Primary Completion 2027-08-31 (Estimated); Study Completion 2027-08-31 (Estimated)

PRIMARY OUTCOMES:
Detection of Actionable Genomic Alterations by ctDNA Profiling | Baseline (within 30 days prior to initiation of systemic therapy or prior to subsequent treatment)
  Frequency of targetable genetic alterations, especially FGFR2 fusion, detected in ctDNA from patients with advanced biliary tract cancer.

SECONDARY OUTCOMES:
Frequency of Specific Genomic Alterations by ctDNA Analysis | Up to 24 months
  Assessment of the frequency of specific genetic alterations (e.g., FGFR2 fusion) identified by ctDNA in Korean patients with advanced biliary tract cancer.
Proportion of Patients Receiving Targeted Therapy Based on ctDNA Findings | Up to 24 months
  Percentage of patients who received targeted therapies (including pemigatinib for FGFR2 fusion) according to ctDNA-based genomic profiling results.

OTHER OUTCOMES:
Association of ctDNA Variant Allele Frequency With Clinical Prognosis | Up to 24 months
  Correlation of maximum variant allele frequency (max VAF) in ctDNA with survival outcomes in advanced biliary tract cancer patients.
Clinical Outcomes in Patients Treated With Targeted Therapy | Up to 24 months
  Proportion of patients achieving complete response, partial response, or stable disease based on RECIST v1.1 criteria among those treated with pemigatinib or other targeted therapies.
Survival Outcomes in Patients Receiving Targeted Therapy | Up to 24 months
  Progression-free survival (PFS) and overall survival (OS) of patients treated with pemigatinib or other targeted therapies according to ctDNA findings.
Resistance Mechanisms and Clonal Evolution Identified by Serial ctDNA Analysis | At progression or up to 24 months
  Exploration of acquired resistance mechanisms and clonal evolution through repeat ctDNA analysis in patients treated with FGFR2 inhibitors such as pemigatinib.
Concordance of Genomic Alterations Between ctDNA and Tissue next-generation sequencing (NGS) | Baseline and up to 24 months
  Assessment of concordance between genomic alterations, including FGFR2 fusion and other actionable mutations, identified by ctDNA and those detected by tissue next-generation sequencing when available.

CONTACTS AND LOCATIONS:
Overall Officials: Hong Jae Chon, Principal Investigator — Principal Investigator
Locations (1):
- CHA Bundang Medical Center, Seongnam-si, Gyeonggi-do, South Korea

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Baria K, De Toni EN, Yu B, Jiang Z, Kabadi SM, Malvezzi M. Worldwide Incidence and Mortality of Biliary Tract Cancer. Gastro Hep Adv. 2022 Apr 15;1(4):618-626. doi: 10.1016/j.gastha.2022.04.007. eCollection 2022. PMID 39132071
- [Background] Valle J, Wasan H, Palmer DH, Cunningham D, Anthoney A, Maraveyas A, Madhusudan S, Iveson T, Hughes S, Pereira SP, Roughton M, Bridgewater J; ABC-02 Trial Investigators. Cisplatin plus gemcitabine versus gemcitabine for biliary tract cancer. N Engl J Med. 2010 Apr 8;362(14):1273-81. doi: 10.1056/NEJMoa0908721. PMID 20375404
- [Background] Oh DY, Ruth He A, Qin S, Chen LT, Okusaka T, Vogel A, Kim JW, Suksombooncharoen T, Ah Lee M, Kitano M, Burris H, Bouattour M, Tanasanvimon S, McNamara MG, Zaucha R, Avallone A, Tan B, Cundom J, Lee CK, Takahashi H, Ikeda M, Chen JS, Wang J, Makowsky M, Rokutanda N, He P, Kurland JF, Cohen G, Valle JW. Durvalumab plus Gemcitabine and Cisplatin in Advanced Biliary Tract Cancer. NEJM Evid. 2022 Aug;1(8):EVIDoa2200015. doi: 10.1056/EVIDoa2200015. Epub 2022 Jun 1. PMID 38319896
- [Background] Valle JW, Lamarca A, Goyal L, Barriuso J, Zhu AX. New Horizons for Precision Medicine in Biliary Tract Cancers. Cancer Discov. 2017 Sep;7(9):943-962. doi: 10.1158/2159-8290.CD-17-0245. Epub 2017 Aug 17. PMID 28818953
- [Background] Abou-Alfa GK, Sahai V, Hollebecque A, Vaccaro G, Melisi D, Al-Rajabi R, Paulson AS, Borad MJ, Gallinson D, Murphy AG, Oh DY, Dotan E, Catenacci DV, Van Cutsem E, Ji T, Lihou CF, Zhen H, Feliz L, Vogel A. Pemigatinib for previously treated, locally advanced or metastatic cholangiocarcinoma: a multicentre, open-label, phase 2 study. Lancet Oncol. 2020 May;21(5):671-684. doi: 10.1016/S1470-2045(20)30109-1. Epub 2020 Mar 20. PMID 32203698
- [Background] Javle M, Roychowdhury S, Kelley RK, Sadeghi S, Macarulla T, Weiss KH, Waldschmidt DT, Goyal L, Borbath I, El-Khoueiry A, Borad MJ, Yong WP, Philip PA, Bitzer M, Tanasanvimon S, Li A, Pande A, Soifer HS, Shepherd SP, Moran S, Zhu AX, Bekaii-Saab TS, Abou-Alfa GK. Infigratinib (BGJ398) in previously treated patients with advanced or metastatic cholangiocarcinoma with FGFR2 fusions or rearrangements: mature results from a multicentre, open-label, single-arm, phase 2 study. Lancet Gastroenterol Hepatol. 2021 Oct;6(10):803-815. doi: 10.1016/S2468-1253(21)00196-5. Epub 2021 Aug 3. PMID 34358484
- [Background] Javle M, Borad MJ, Azad NS, Kurzrock R, Abou-Alfa GK, George B, Hainsworth J, Meric-Bernstam F, Swanton C, Sweeney CJ, Friedman CF, Bose R, Spigel DR, Wang Y, Levy J, Schulze K, Cuchelkar V, Patel A, Burris H. Pertuzumab and trastuzumab for HER2-positive, metastatic biliary tract cancer (MyPathway): a multicentre, open-label, phase 2a, multiple basket study. Lancet Oncol. 2021 Sep;22(9):1290-1300. doi: 10.1016/S1470-2045(21)00336-3. Epub 2021 Jul 30. PMID 34339623
- [Background] Abou-Alfa GK, Macarulla T, Javle MM, Kelley RK, Lubner SJ, Adeva J, Cleary JM, Catenacci DV, Borad MJ, Bridgewater J, Harris WP, Murphy AG, Oh DY, Whisenant J, Lowery MA, Goyal L, Shroff RT, El-Khoueiry AB, Fan B, Wu B, Chamberlain CX, Jiang L, Gliser C, Pandya SS, Valle JW, Zhu AX. Ivosidenib in IDH1-mutant, chemotherapy-refractory cholangiocarcinoma (ClarIDHy): a multicentre, randomised, double-blind, placebo-controlled, phase 3 study. Lancet Oncol. 2020 Jun;21(6):796-807. doi: 10.1016/S1470-2045(20)30157-1. Epub 2020 May 13. PMID 32416072
- [Background] Zhu AX, Macarulla T, Javle MM, Kelley RK, Lubner SJ, Adeva J, Cleary JM, Catenacci DVT, Borad MJ, Bridgewater JA, Harris WP, Murphy AG, Oh DY, Whisenant JR, Lowery MA, Goyal L, Shroff RT, El-Khoueiry AB, Chamberlain CX, Aguado-Fraile E, Choe S, Wu B, Liu H, Gliser C, Pandya SS, Valle JW, Abou-Alfa GK. Final Overall Survival Efficacy Results of Ivosidenib for Patients With Advanced Cholangiocarcinoma With IDH1 Mutation: The Phase 3 Randomized Clinical ClarIDHy Trial. JAMA Oncol. 2021 Nov 1;7(11):1669-1677. doi: 10.1001/jamaoncol.2021.3836. PMID 34554208
- [Background] Le DT, Kim TW, Van Cutsem E, Geva R, Jager D, Hara H, Burge M, O'Neil B, Kavan P, Yoshino T, Guimbaud R, Taniguchi H, Elez E, Al-Batran SE, Boland PM, Crocenzi T, Atreya CE, Cui Y, Dai T, Marinello P, Diaz LA Jr, Andre T. Phase II Open-Label Study of Pembrolizumab in Treatment-Refractory, Microsatellite Instability-High/Mismatch Repair-Deficient Metastatic Colorectal Cancer: KEYNOTE-164. J Clin Oncol. 2020 Jan 1;38(1):11-19. doi: 10.1200/JCO.19.02107. Epub 2019 Nov 14. PMID 31725351
- [Background] Lamarca A, Kapacee Z, Breeze M, Bell C, Belcher D, Staiger H, Taylor C, McNamara MG, Hubner RA, Valle JW. Molecular Profiling in Daily Clinical Practice: Practicalities in Advanced Cholangiocarcinoma and Other Biliary Tract Cancers. J Clin Med. 2020 Sep 3;9(9):2854. doi: 10.3390/jcm9092854. PMID 32899345
- [Background] Strickler JH, Loree JM, Ahronian LG, Parikh AR, Niedzwiecki D, Pereira AAL, McKinney M, Korn WM, Atreya CE, Banks KC, Nagy RJ, Meric-Bernstam F, Lanman RB, Talasaz A, Tsigelny IF, Corcoran RB, Kopetz S. Genomic Landscape of Cell-Free DNA in Patients with Colorectal Cancer. Cancer Discov. 2018 Feb;8(2):164-173. doi: 10.1158/2159-8290.CD-17-1009. Epub 2017 Dec 1. PMID 29196463
- [Background] Goyal L, Saha SK, Liu LY, Siravegna G, Leshchiner I, Ahronian LG, Lennerz JK, Vu P, Deshpande V, Kambadakone A, Mussolin B, Reyes S, Henderson L, Sun JE, Van Seventer EE, Gurski JM Jr, Baltschukat S, Schacher-Engstler B, Barys L, Stamm C, Furet P, Ryan DP, Stone JR, Iafrate AJ, Getz G, Porta DG, Tiedt R, Bardelli A, Juric D, Corcoran RB, Bardeesy N, Zhu AX. Polyclonal Secondary FGFR2 Mutations Drive Acquired Resistance to FGFR Inhibition in Patients with FGFR2 Fusion-Positive Cholangiocarcinoma. Cancer Discov. 2017 Mar;7(3):252-263. doi: 10.1158/2159-8290.CD-16-1000. Epub 2016 Dec 29. PMID 28034880
- [Background] Miller AM, Shah RH, Pentsova EI, Pourmaleki M, Briggs S, Distefano N, Zheng Y, Skakodub A, Mehta SA, Campos C, Hsieh WY, Selcuklu SD, Ling L, Meng F, Jing X, Samoila A, Bale TA, Tsui DWY, Grommes C, Viale A, Souweidane MM, Tabar V, Brennan CW, Reiner AS, Rosenblum M, Panageas KS, DeAngelis LM, Young RJ, Berger MF, Mellinghoff IK. Tracking tumour evolution in glioma through liquid biopsies of cerebrospinal fluid. Nature. 2019 Jan;565(7741):654-658. doi: 10.1038/s41586-019-0882-3. Epub 2019 Jan 23. PMID 30675060
- [Background] Hwang S, Woo S, Kang B, Kang H, Kim JS, Lee SH, Kwon CI, Kyung DS, Kim HP, Kim G, Kim C, Chon HJ. Concordance of ctDNA and tissue genomic profiling in advanced biliary tract cancer. J Hepatol. 2025 Apr;82(4):649-657. doi: 10.1016/j.jhep.2024.10.020. Epub 2024 Oct 21. PMID 39442892
- [Background] Berchuck JE, Facchinetti F, DiToro DF, Baiev I, Majeed U, Reyes S, Chen C, Zhang K, Sharman R, Uson Junior PLS, Maurer J, Shroff RT, Pritchard CC, Wu MJ, Catenacci DVT, Javle M, Friboulet L, Hollebecque A, Bardeesy N, Zhu AX, Lennerz JK, Tan B, Borad M, Parikh AR, Kiedrowski LA, Kelley RK, Mody K, Juric D, Goyal L. The clinical landscape of cell-free DNA alterations in 1671 patients with advanced biliary tract cancer. Ann Oncol. 2022 Dec;33(12):1269-1283. doi: 10.1016/j.annonc.2022.09.150. Epub 2022 Sep 9. PMID 36089135
- [Background] Ettrich TJ, Schwerdel D, Dolnik A, Beuter F, Blatte TJ, Schmidt SA, Stanescu-Siegmund N, Steinacker J, Marienfeld R, Kleger A, Bullinger L, Seufferlein T, Berger AW. Genotyping of circulating tumor DNA in cholangiocarcinoma reveals diagnostic and prognostic information. Sci Rep. 2019 Sep 13;9(1):13261. doi: 10.1038/s41598-019-49860-0. PMID 31519967
- [Background] Goyal L, Shi L, Liu LY, Fece de la Cruz F, Lennerz JK, Raghavan S, Leschiner I, Elagina L, Siravegna G, Ng RWS, Vu P, Patra KC, Saha SK, Uppot RN, Arellano R, Reyes S, Sagara T, Otsuki S, Nadres B, Shahzade HA, Dey-Guha I, Fetter IJ, Baiev I, Van Seventer EE, Murphy JE, Ferrone CR, Tanabe KK, Deshpande V, Harding JJ, Yaeger R, Kelley RK, Bardelli A, Iafrate AJ, Hahn WC, Benes CH, Ting DT, Hirai H, Getz G, Juric D, Zhu AX, Corcoran RB, Bardeesy N. TAS-120 Overcomes Resistance to ATP-Competitive FGFR Inhibitors in Patients with FGFR2 Fusion-Positive Intrahepatic Cholangiocarcinoma. Cancer Discov. 2019 Aug;9(8):1064-1079. doi: 10.1158/2159-8290.CD-19-0182. Epub 2019 May 20. PMID 31109923
- [Background] Chae H, Kim D, Yoo C, Kim KP, Jeong JH, Chang HM, Lee SS, Park DH, Song TJ, Hwang S, Kim KH, Song GW, Ahn CS, Lee JH, Hwang DW, Kim SC, Jang SJ, Hong SM, Kim TW, Ryoo BY. Therapeutic relevance of targeted sequencing in management of patients with advanced biliary tract cancer: DNA damage repair gene mutations as a predictive biomarker. Eur J Cancer. 2019 Oct;120:31-39. doi: 10.1016/j.ejca.2019.07.022. Epub 2019 Aug 30. PMID 31476489
- [Background] Awosika JA, Monge C, Greten TF. Integration of circulating tumor DNA in biliary tract cancer: the emerging landscape. Hepat Oncol. 2024 Dec 31;11(1):2403334. doi: 10.1080/20450923.2024.2403334. Epub 2024 Oct 9. PMID 39881555